CLINICAL TRIAL: NCT07170683
Title: An Investigation of Microperimetry for Monitoring Retinal Function in Selected Macular Disorders
Brief Title: Microperimetry Changes in Retinal Function in Macular Disorders
Acronym: MAIAStud
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 24060
Record Dates: First submitted 2025-07-08; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Dry AMD; Diabetic Retinopathy (DR)
Keywords: retinal sensitivity; microperimetry; diabetic retinopathy; dry AMD; OCT; OCT-A; geographic atrophy
MeSH Terms: conditions — Diabetic Retinopathy; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with dry AMD (including geographic atrophy [GA]): Participants with dry AMD including GA. MP will be performed in 2 different modalities, a full staircase threshold stimuli projection, and a simplified stimuli projection of 4 fixed levels of stimuli intensity.
  OCT and OCT-A will be done with the Topcon Triton. Best habitual corrected distance VA (logMAR) will be recorded.
  Interventions: Other: MAIA Microperimetry; Device: Microperimetry; Other: Visual Acuity Measurement (logMAR); Device: OCT-A
- Persons with diabetes without diabetic retinopathy: Participants with diabetes without diabetic retinopathy. MP will be performed in 2 different modalities, a full staircase threshold stimuli projection, and a simplified stimuli projection of 4 fixed levels of stimuli intensity.
  OCT and OCT-A will be done with the Topcon Triton. Best habitual corrected distance VA (logMAR) will be recorded.
  Interventions: Other: MAIA Microperimetry; Device: Microperimetry; Other: Visual Acuity Measurement (logMAR); Device: OCT-A
- Participants with diabetes with mild to moderate diabetic retinopathy (i.e. non-proliferative DR)..: Participants with diabetes with mild to moderate diabetic retinopathy. MP will be performed in 2 different modalities, a full staircase threshold stimuli projection, and a simplified stimuli projection of 4 fixed levels of stimuli intensity.
  OCT and OCT-A will be done with the Topcon Triton. Best habitual corrected distance VA (logMAR) will be recorded.
  Interventions: Other: MAIA Microperimetry; Device: Microperimetry; Other: Visual Acuity Measurement (logMAR); Device: OCT-A
- Normal (healthy) controls: Normal controls will include persons who are not diabetic, and do not have glaucoma, any retinal or optic nerve disease.
  MP will be performed in 2 different modalities, a full staircase threshold stimuli projection, and a simplified stimuli projection of 4 fixed levels of stimuli intensity.
  OCT and OCT-A will be done with the Topcon Triton. Best habitual corrected distance VA (logMAR) will be recorded.
  Interventions: Other: MAIA Microperimetry; Device: Microperimetry; Other: Visual Acuity Measurement (logMAR); Device: OCT-A

INTERVENTIONS:
Other: MAIA Microperimetry — Microperimetry (MP) is not performed as part of the current NHS patient pathway. We plan testing 2 MP strategies ('standard' vrs 'fast') to determine whether the fast testing strategy is as robust as the standard test strategy. Adopting the fast strategy will reduce time spent on the MP machine to obtain relevant test results. Healthy volunteers (with no retinal disease) are necessary for comparison, and to establish validity of any new findings.
Device: Microperimetry — Two fully automatic MAIA MP (CenterVue, spa; Padova, Italy) examinations (to obtain retinal sensitivity) shall be performed over the 10° diameter central retinal area for the recruited study participants. The first one will be performed with a fast projection, and the second one with the standard full 4-2 staircase projection strategy. Identification of the PRL area will be automatically calculated at the end of each examination. All patient groups will have identical assessment, at all time points. Healthy volunteers will only have assessments at baseline (one examination only)..
Other: Visual Acuity Measurement (logMAR) — Visual acuity will be measured with the ETDRS chart, and with the participant habitual distance correction, and recorded in logMAR notation
Device: OCT-A — OCT and OCT-A examination, as well FAF will be undertaken with the Topcon Triton Plus OCT

SUMMARY:
The purpose of this study is to measure precisely how sensitive the central part of the retina - the light-sensitive film at the back of the eye, is to light. We will use a special device called the Macular Integrity Assessment (MAIA) microperimetry (MP) system to achieve this, particularly for individuals with specific retinal conditions. The macula (with the fovea at its very centre) is the part of the retina responsible for our fine detailed vision, colour vision, and maintaining steady gaze on objects (called 'fixation'). Diseases that affect the macula lead to difficulties in seeing clearly.

Macular sensitivity refers to how responsive the macula is to light, including the ability to read and focus on objects. This also determines how well the eye can maintain a steady gaze on objects of interest ('fixation'). While standard eye tests primarily measure vision in the fovea, measuring sensitivity across the wider macula would provide a more complete picture of visual function. Furthermore, we believe that macular sensitivity changes are often one of the earliest signs of retinal diseases, before a person experiences blurry vision. Currently, MP is not used routinely in UK NHS clinical practice.

The commonest retinal diseases are age-related macular degeneration (AMD) and diabetic retinopathy (DR). There are 2 types of AMD: dry and wet.

* Dry AMD is a condition that affects the central part of the retina (the macula) and can lead to gradual vision loss as people age. This is due to wearing out and loss of the slight sensitive cells in the macula that can make it harder to see fine details, such as reading or recognizing faces.
* Diabetic retinopathy means that diabetes has affected the blood vessels in the retina. In the early stages, the affected blood vessels do not leak. However, progression results in leakage of the blood vessels in the retina, leading to retinal swelling (called diabetic macular oedema [DMO]). Eyes with DMO function less well compared to when there is no swelling.

It is important to investigate these selected common conditions further, in order to find ways of detecting changes earlier, before the patient notices any abnormalities. Such earlier detection may result in better understanding and treatments in the future.

The main goal of this research is to measure macular sensitivity and ability to maintain a steady gaze on specific objects or points in patients with these macular disorders using the MAIA device. These measurements will be compared to changes in the structure of the macula, obtained using advanced imaging techniques like optical coherence tomography (OCT) and OCT angiography (OCTA), which are routinely used in standard clinical practice.

This study will form part of a research/educational thesis, and provide additional data to complement previous research on the topic.

Participants (after consent) will have MP done. In addition, we will assess information from their eye clinic records, including images and scans of the back of the eyes (OCT and OCTA). No treatment interventions are planned as part of this study. Participants standard of care will not be affected.

Participants will have tests done at baseline, and repeated at 6 and 12 months. In addition, we will invite a group of normal controls (i.e. persons who do not have any diseases of the back of their eyes) for comparison. This will ensure validity of our findings. The normal controls will attend only once (at baseline). After consent is obtained, these healthy participants will have MP, and imaging of the macula with OCT.

ELIGIBILITY:
A. Patients

Inclusion Criteria:

* Adult age above 21 years old.
* Signed informed consent
* Visual acuity Log MAR 0.0 to 1.2
* Patients diagnosed with:

  * Geographic atrophy (AMD).
  * Diabetic without retinopathy, and minimal to moderate non-proliferative diabetic retinopathy (NPDR) with or without presence of macular oedema on optical coherence tomography (OCT)
* Control group of age matched participants without any retinal disease, glaucoma or optic nerve disease in either eye Patients willing to attend follow-up MP examinations. (This does not apply to normal controls who only require one attendance).

Exclusion Criteria

* Moderate to severe cataract (over grade 2) or other cause of opaque optical media that will preclude adequate fundoscopy or MP assessment.
* Previous treatments in the eye with intravitreal therapies of anti-VEGFs or steroids within the previous 6 months, or macular laser photocoagulation
* Active vascular event in either eye any examination time.
* Participants who are unable/unwilling to provide consent
* Participants who are unable to read English fluently

B. Normal Controls Inclusion Criteria

* Normal controls will include persons who are not diabetic, and do not have glaucoma, any retinal or optic nerve disease.
* Signed informed consent
* Adult age above 21 years old. No upper age limit.
* Visual acuity LogMAR <0.2.
* Controls should be willing to attend once only.

Exclusion criteria

* Moderate to severe cataract (over grade 2) or other cause of opaque optical media
* Previous treatments in the particular eye with intravitreal therapies of anti-VEGFs or steroids within the previous 6 months, or macular laser photocoagulation
* Active/previous vascular event in either eye e.g. retinal arterial or vein occlusion, ischaemic optic neuropathy, or glaucoma
* Persons with diabetes
* Participants who are unable to read English fluently
* Participants who are unable/unwilling to provide consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Medical Retina and Macular clinics of the Queen's Medical Centre.
  Healthy controls will be recruited from persons accompanying patients to the Eye Clinic, hospital and University staff. Healthy volunteers who are accompanying persons to the clinic will be approached after the patient participant has been approached.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Correlations of retinal sensitivity (dB) changes over time, compared with OCT/OCTA measures (change in retinal/choroidal thickness in microns and/or %; % change in choroidal vascularity) | from enrolment (baseline) to 6 and 12 months
  Retinal sensitivity (dB) will be measured with MP. Correlations will be made between retinal sensitivities between each group and normal controls, and over time.
MP BCEA values | Baseline compared to 6 and 12 months
  Correlations of changes in BCEA (fixation stability in degrees: BCEA@63 and BCEA@95) in the different groups will be analysed similarly, and over time, using a mixed-effects model to account for variability between eyes and between subjects. Quantify deviations from baseline PRL in degrees.

SECONDARY OUTCOMES:
Baseline factors relationship to retinal sensitivity (dB) with age (years), disease duration (years) and baseline visual acuity (LogMAR) | baseline, changes from baseline to 6 and 12 months
  Relationship of baseline factors (e.g., age [years], disease duration [years], baseline visual acuity [logMAR]) are predictive of outcomes in retinal sensitivity (dB), fixation stability (BCEA), or fixation (PRL) location. Statistical correlations will be made of retinal sensitivities (dB) between each group(dry AMD, no DR, DR) and normal controls, and over time

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No